CLINICAL TRIAL: NCT01740778
Title: Lancing Device Comparison Study
Status: Completed | Type: Observational
Sponsor: Facet Technologies (Other)
Responsible Party: Principal Investigator, Mary Kate Pynes, CRA, Facet Technologies
Other Study IDs: FT-2009-Aurora
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; Medical Device; Lancing
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Study Group 1: Aurora vs. Microlet 2
- Study Group 2: Aurora vs. SoftClix
- Study Group 3: Aurora vs. One Touch Comfort
- Study Group 4: Aurora vs. Multiclix

SUMMARY:
To evaluate pain responses using the Aurora lancing device and Velvet 33g lancet compared to other common, commercially available lancing systems. Subjects will test the devices at a depth setting sufficient to provide enough blood volume to trigger the OneTouch® Ultra®Mini blood glucose meter using OneTouch® Ultra® blood glucose test strips from either the fingertip or alternate site testing.

DETAILED DESCRIPTION:
A low-pain lancing is being developed code name Aurora) for use with a 33g proprietary lancet (code name Velvet). This study evaluates the pain associated with finger lancing using this device and compares that pain to other commercially available lancing devices and associated lancets.

All lancets used in the study are currently commercially available except the Facet 33g lancet, which is a prototype version of commercially available lancets.

The Roche Multiclix, Roche Softclix, One Touch Comfort and Bayer Microlet 2 lancing devices are all commercially available.

The Aurora Lancing Device is effective in obtaining a sufficient blood sample for performing an accurate blood glucose measurement; and the benefits of using the Aurora Lancing Device outweighs any residual risks associated with the product. Literature concerning blood glucose testing was researched by using popular medical databases such as pubmed.gov, diabeteshealth.com, clinicaltrial.gov and search terms lancing device, clinical study, blood volume and pain. Using other popular search engines such as Google was beneficial in helping to support claims concerning safety and efficacy. A commercial database company, NERAC was used as a part of the literature research effort. Our review, together with preliminary in-house bench testing, shows that the Aurora Lancing Device should be able to:

* Obtain enough blood volume for a meter reading that measures blood glucose levels;
* Is as safe as comparative lancing devices currently on the market;
* Produces no more pain than comparative lancing devices currently on the market using a 28 gauge needle; and
* Is representative of "current state of the art" The Aurora Lancing Device uses a 33 gauge, uniquely designed lancet developed under project Velvet. The blood lancet is designed so that it can only be used in the Aurora lancing device. The lancing device features multiple depth settings and includes alternate site test capability. The lancet guidance system is designed to maximize lancet control thereby increasing comfort and reducing pain perception. The Aurora lancing device is comparable to the Roche Softclix and other lancing devices already in commercial distribution. Like Aurora the Roche Softclix lancing device offers diabetics a unique lancet design and precise lancet motion. Roche Softclix uses a 28 gauge lancet and has eleven depth settings as well as alternative site test capability.

ELIGIBILITY:
Inclusion Criteria:

Must have been diagnosed with type 1 or type 2 diabetes for at least 1 year Must be doing SMBG, at least twice daily for at least 6 months Must be 18 years of age and older Must have healthy fingers and hands Must be able to read instructions in English. Must be able to perform all tasks in the protocol.

Exclusion Criteria:

Subjects with neuropathy or any other nerve damage in the hand or fingers (this will be discovered through the monofilament test)

Subjects who are taking prescription anti-coagulants or more than one full aspirin per day during the past week or have clotting problems that may prolong bleeding (persons taking Plavix or a daily low dose aspirin will not be excluded but this will be recorded).

Subjects taking prescription medications for neuropathy.

Subjects with hemophilia or any other bleeding disorder.

subjects with infection with a blood borne pathogen (e.g., HIV, hepatitis).

Subjects having a condition such as a cognitive disorder, which in the opinion of the Investigator would put the person at risk or seriously compromise the integrity of the study (PI will sign CRF if subject is excluded).

Subjects with missing digits.

Subjects who are pregnant or nursing.

Subjects on chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gender: Approximately 50% male, 50% female; Type Diabetes: 25% Type 1, 75% Type 2 Age: 18 or older
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Reading | 1-1 hour visit during the study
  During the first part of the study, subjects will test their lancing devices at a depth setting sufficient to provide enough blood volume to trigger the OneTouch® Ultra®Mini blood glucose meter using OneTouch® Ultra® blood glucose test strips.
  The second part of the study will generate the pain data associated with the Alternate site testing (AST) will also be performed on the palm of the hand and the forearm with the Aurora device and Velvet 33g lancet.
  Each lancing event, in the first portion of the study, is considered successful if at least 2 out of 3 lancing events are successful in producing enough blood to trigger the One Touch® Ultra®Mini blood glucose meter.

SECONDARY OUTCOMES:
Pain Scale Rating | 1- 1 hour visit during the study
  The second part of the study will generate the pain data associated with the Aurora device and Velvet 33g lancet along with the study comparative device. During the second visit, alternate site testing (AST) will also be performed on the palm of the hand and the forearm with the Aurora device and Velvet 33g lancet.
  The second portion of the study will compare and report the differences in pain between the device/lancet combinations. Pain will be assessed for each successful fingerstick per the visual analog scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shemain, MBA, Principal Investigator — SHEMAIN CONSULTING GROUP, LLC